CLINICAL TRIAL: NCT04436861
Title: Demonstration of the Level of Anxiety / Depression of Healthcare Professionals and Non-healthcare Professionals One Month After the Confinement Period
Brief Title: the Health Crisis at the Healthcare Professionals, Careers and Non-careers, a Month After the Containment Period
Status: Withdrawn | Type: Observational
Why Stopped: the sponsor decided to stop the study
Sponsor: Clinique Medipole Garonne (Other)
Responsible Party: Sponsor
Other Study IDs: Decovid
Record Dates: First submitted 2020-06-11; First posted 2020-06-18 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-04

CONDITIONS: Psychology, Social

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigator wish to study, at a distance from the lifting of confinement (1 month), whether the psychological impact on professionals in nursing and non-nursing care establishments is associated with their living context (professional and personal situation) during confinement.

DETAILED DESCRIPTION:
The context of confinement and of the global pandemic is a major source of stress for the entire population: separation of loved ones, loss of freedom, uncertainty about the infectious status, boredom. All of these factors can cause negative mental health consequences. Having little social contact was one of the factors increasing the negative psychological impact of confinement.

People suffering from psychological disorders are particularly vulnerable during quarantine periods. On March 17, 2020, the French government implemented national containment measures due to the Covid-19 epidemic.

Although the effects of containment have been studied for fragile populations, no study to date has focused on the specific population of healthcare facility staff. These caregivers have for the most part continued their professional activity, but they have been confronted with the fear of contracting or causing patients to contract Covid-19.

At a distance from the lifting of confinement (1 month), the investigator wish to study whether the highlighting of anxiety or depression in these healthcare professionals is associated with their context of life (professional and personal situation) during confinement

ELIGIBILITY:
Inclusion Criteria:

* Nursing and non-nursing care professionals

Exclusion Criteria:

* Refusal to participate
* Subject included in an interventional study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We are not basing the study size on statistical arguments for this observational study. The study will be offered to all healthcare professionals in order to limit bias. However, we expect a minimum of 200 responses
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-28 (Actual); Primary Completion 2020-06-28 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Demonstration of the level of anxiety / depression of healthcare professionals and non-healthcare professionals one month after the confinement period | 1 month
  Anxiety-depression will be assessed by the hospital anxiety and depression scalequestionnaire. The context of life during confinement will be assessed by a self-questionnaire collecting data relating to lifestyle and work.

IPD SHARING:
Plan to Share IPD: No